CLINICAL TRIAL: NCT06063915
Title: "Efficacy of Isoinertial Rehabilitation in Recovering Hamstring Strength Following Surgical Anterior Cruciate Ligament Reconstruction: a Randomized Controlled Trial"
Brief Title: Isoinertial Rehabilitation in Recovering Hamstring Strength Following Surgical Anterior Cruciate Ligament Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli studi di Roma Foro Italico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISOHAMACL
Record Dates: First submitted 2023-07-28; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: ACL Injury; ACL Sprain; ACL Tear; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gold Rehab + Strength Training (Active Comparator): Gold standard rehabilitation plus traditional strength training with overloads
  Interventions: Other: Strength Training
- Gold Rehab + Isoinertial (Experimental): Gold standard rehabilitation with the inclusion of isoinertial training
  Interventions: Device: Isoinertial training

INTERVENTIONS:
Device: Isoinertial training — The subjects included in the study will undergo traditional muscle strengthening for a period of 4 weeks, with 2 sessions per week consisting of strength training using isoinertial machines
  Arms: Gold Rehab + Isoinertial
Other: Strength Training — The subjects included in the study will undergo traditional muscle strengthening for a period of 4 weeks, with 2 sessions per week consisting of strength training using classic exercises
  Arms: Gold Rehab + Strength Training

SUMMARY:
The present experimental study aims to evaluate the effectiveness and tolerability of isoinertial strength training of the hamstrings using machines in patients with ACL-R during the intermediate post-intervention phases.

DETAILED DESCRIPTION:
A proper post-operative rehabilitation program is essential for a positive outcome after anterior cruciate ligament (ACL) reconstruction surgery, a procedure known to cause morpho-functional issues in the short, medium, and long term in individuals who undergo it. Generally, after an initial rehabilitation phase focused on protecting the healing process of the new ligament and regaining range of motion, the rehabilitation path focuses on muscular strengthening and neuromuscular control of both lower limbs. It has been demonstrated that deficits in extensor and flexor muscle strength, as well as their strength ratios, increase the risk of re-injury. Specifically, in athletes, the rate of recurrence, defined as a new injury to the same or opposite side ACL, is considerably high.

High-intensity resistance training of the operated limb has often been contraindicated in the early post-operative period, as it was considered detrimental to the new ligament, joint cartilage, and surrounding soft tissues. However, recent studies suggest that the early application of progressive eccentric-focused exercises, even with high loads, can be safely used to increase muscle volume and strength levels in individuals undergoing ACL reconstruction (ACL-R). Therefore, eccentric reinforcement can be a valid alternative to traditional concentric work for improving lower limb muscle strength after ACL-R.

Recently, it has been demonstrated that strength training using isoinertial machines in healthy individuals leads to positive chronic adaptations in terms of strength recovery, power, and functional capacities such as sprinting, change of direction, and agility. Isoinertial training allows for exercises in both closed and open kinetic chains, as well as multiplanar motor activities. The combination of concentric phases with subsequent eccentric overload allows for the development of high levels of strength and power with low energy cost, promotes intermuscular coordination, preferentially recruits motor units with high activation thresholds, and increases cortical activity. Increased muscle activation, particularly during eccentric muscle actions, indicates a higher mechanical load and a greater training stimulus, leading to better and earlier protein synthesis and subsequent muscle hypertrophy compared to traditional resistance training. Furthermore, the metabolic cost required for an eccentric contraction is about a quarter of that for a concentric contraction at the same external load. Therefore, at the same contraction velocity, eccentric contractions allow for a higher force expression.

While the use of isoinertial equipment is well-established in healthy individuals, scientific evidence regarding its use in rehabilitation protocols is currently limited. The use of eccentric overload, in addition to improving parameters related to muscle strength and power, seems to promote tendon remodeling due to an increased production of fibroblasts and collagen, generated by the higher mechanical load compared to traditional concentric exercise. In lower limb pathologies, isoinertial rehabilitation following injury can be a valid alternative to traditional strength training for the development of muscle hypertrophy and function. However, specific studies investigating the effects of isoinertial rehabilitation in the intermediate stages of recovery following ACL-R and monitoring the tolerability of the treatment are currently lacking.

ELIGIBILITY:
Inclusion Criteria:

* having undergone ACL-R surgery following a unilateral rupture
* with reconstructive surgical technique using autograft tendon from the semitendinosus and gracilis muscles (ST-GR), also in the presence of meniscal injuries treated with selective meniscectomy or meniscal suturing.
* Participants must report a level of physical activity between 5 and 10 assessed using the Tegner scale, and have completed the third month of post-operative rehabilitation

Exclusion Criteria:

* concurrent injuries involving other ligaments of the knee, cartilage injuries requiring surgery to repair the damage
* previous ACL reconstruction (re-rupture with a new ACL reconstruction) on the knee affected by the new ACL injury.
* Additionally, if the level of pain prevents the subject from performing the functional tests, they will not be included in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Active and passive range of motion (ROM) of the knee joint | Day 0
Active and passive range of motion (ROM) of the knee joint | Day 28
Strength of the thigh flexor and extensor muscles | Day 0
Strength of the thigh flexor and extensor muscles | Day 28
Qualitative analysis of the Single Leg Squat | Day 0
Qualitative analysis of the Single Leg Squat | Day 28
Maximal Hip Flexion Active Knee Extension Test | Day 0
Maximal Hip Flexion Active Knee Extension Test | Day 28
Quantitative analysis of the Drop Jump, with frontal and sagittal views | Day 0
Quantitative analysis of the Drop Jump, with frontal and sagittal views | Day 28

IPD SHARING:
Plan to Share IPD: Undecided